CLINICAL TRIAL: NCT04489485
Title: Online System for Identifying and Addressing Teen Depression in Primary Care
Acronym: Depression
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Total Child Health, Inc. (Industry)
Collaborators: National Institute of Mental Health (NIMH) (NIH); Foresight Logic (Other)
Responsible Party: Principal Investigator, Barbara Howard, MD, President of Total Child Health, Total Child Health, Inc.
Other Study IDs: R44MH116751 (NIH); 1R44MH116751-01A1 (NIH)
Record Dates: First submitted 2020-06-19; First posted 2020-07-28 (Actual); Last update posted 2022-03-22 (Actual); Status verified 2022-03

CONDITIONS: Major Depression; Dysthymia; Depressive Symptoms
Keywords: depression
MeSH Terms: conditions — Depressive Disorder, Major; Dysthymic Disorder; Depression

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (5):
- Primary Care Providers (PCP): 20 PCP who provide well child care to teens 12-18. After randomization, 10 PCPs in the enhanced care group will use the Teen Depression Module for care.
  Interventions: Behavioral: Teen Depression Module used for care
- Standard care teens: All teens coming for routine well child care to the control group PCPs will have routine depression screening and Youth Health Questionnaire without goals to inform treatment as usual. They will be offered a goals text messaging conversation. Suicide screening will be at the discretion of the PCP.
- Enhanced care teens: All teens coming for routine well child care to the enhanced group PCPs will have depression screening with strengths and goals and a depression screen with follow up suggestions for activities to help any depression symptoms, as well as Youth Health Questionnaire with goals and then they will receive treatment guided by the Teen Depression Module and offered a depression text messaging conversation. Suicide screening will be conducted.
  Interventions: Behavioral: Teen Depression Module used for care
- Standard care- caregivers: All caregivers of teens <18 years old coming for routine well child care to the control group PCPs will complete a Pediatric Symptom Checklist and Short Moods and Feelings Questionnaire, plus a Youth Health Questionnaire- Parent version to inform treatment as usual. If the internalizing subscale is positive the caregiver will also complete the Short Moods and Feelings Questionnaire and 3, 6 and 11.5 month follow up report of Intervention received (Parent Intervention Questionnaire)
- Enhanced care- caregivers: All caregivers of teens <18 years old coming for routine well child care to the enhanced group PCPs will complete a Pediatric Symptom Checklist plus a Youth Health Questionnaire- Parent version to inform treatment as usual. If the internalizing subscale is positive the caregiver will also complete the Short Moods and Feelings Questionnaire and 3, 6 and 11.5 month follow up report of Intervention received (Parent Intervention Questionnaire)

INTERVENTIONS:
Behavioral: Teen Depression Module used for care — All teens coming for routine well child care to the enhanced group PCPs will have depression screening with strengths and goals and a depression screen with follow up suggestions for activities to help any depression symptoms, and treatment using the Teen Depression Module and offered a depression chabot. Suicide screening will be conducted.
  Groups: Enhanced care teens; Primary Care Providers (PCP)

SUMMARY:
A novel web-based module (Teen Depression Module or TDM)has been created for assisting primary care providers (PCPs) in screening for and addressing and referring teens with depression. This is a cluster randomized Quality Improvement study to determine if use of the TDM that includes collecting information on strengths and goals as part of well child care will improve detection of depression, referral success, and teen's use of alternative helping strategies with resulting improvement in depression symptoms.

DETAILED DESCRIPTION:
Phase II Summary for finalizing and testing the CHADIS Teen Depression Module (TDM) These aims are unchanged except that health screening visits may be in-person or conducted via telehealth.

II-1. Revise programming and training materials: TDM- an addition for primary care screening and care for teen depression as part of the Comprehensive Health and Decision Information System (CHADIS) online questionnaire delivery system with decision support including "motivational interviewing teleprompters", care coordination functionality for referrals, and text chats- will be revised and programmed as needed to adjust for Phase 1 feedback and training materials created.

II-2 Recruit 20 study PCP's, set up care coordination with MH specialists and assess: Investigators will recruit 20 primary care providers (PCPs), assuring representative Medicaid-insured teens, and randomize to intervention or control. Intervention PCPs will identify their local Mental Health (MH) resources to recruit for referrals and use of care coordination functionality. 2 Therapists, 2 PCPs, and 2 Psychiatrists (Psy) using the care coordination will give feedback on functionality, acceptability and likelihood of continued use as well as use of a text messaging robot messaging about referrals after the baseline. Investigators will document current PCP access to MH services.

II-3 Baseline (3 mo.), refine implementation strategies using QI Maintenance of Certification (MOC-4) sessions:

All 20 PCPs will use the Patient Health Questionnaire-9 (PHQ-9) for depression (without follow-up questions) for a baseline, and have implementation issues addressed using Quality Improvement (QI) methods. Data will be collected from teens and parents before in person or telehealth Health Supervision Visits (HSV) using CHADIS. Data on rates of depression screening using CHADIS and billing data will be shared with PCPs as part of Maintenance of Certification Part 4 (MOC-4) sessions for intervention and controls. Teens (<=480) will be sent a text survey post visit of any strength- or emotion- supporting care received.

II-4 Create child psychiatry version of TDM: Denver team will modify TDM for Psy including care plans.

II-5 Obtain MOC-4 approval for child psychiatry by American Board of Medical Specialties (covering American Board of Psychiatry and Neurology) for Child Psychiatrists for use of the TDM created in II-4 and MOC-4 will be offered to participating Child Psychiatrists.

II-6 Intervention trial: (See Figure) Primary Question 1 (PQ1). For teens PHQ positive, does TDM use result in lower Short Mood & Feelings Questionnaire (SMFQ) scores at 3-, 6-and 11.5-months vs at start of intervention? Primary Question 2. For teens PHQ positive, does TDM use result in lower teen and parent SMFQ scores at 3-, 6-and 11.5-months vs controls? Secondary Question 1 (SQ1): Of teens PHQ positive, does TDM use result in higher rates of accessing treatment at 3-, 6-and 11.5 months vs controls? Secondary Question 2. Does QI method increase rates of teens screened? Secondary Question 3. Does QI method increase rates of Ask Suicide Questions (ASQ) screening? Design: A cluster randomized trial with a 2-group pretest-posttest design clustered at the PCP level will determine pre-post differences within patients and intervention vs control group differences.

Sample size estimates consider the design effect and use an Intent to Treat model. Sample sizes of 107/PCP in both intervention and control will achieve 89.5% power to detect a difference between group means of >=2; also sufficient power for Secondary Questions 1-3. Procedure: Both groups: All teens before HSV will do: Visit Priorities, Teen Health & Goals comprehensive of standard guidelines, and PHQ-9 with follow up to SMFQ, if positive and get health information chats with links to education/advice in their CHADIS Care Portal. All parents will do Visit Priorities and Pediatric Symptom Checklist-17 (PSC) for behavior/mood with follow-up parent SMFQ if the internalizing subscale is positive and can access "handouts" in the parent Care Portal. All PCPs see questionnaire results and earn MOC-4. Intervention group: Teens: will do: goals/strengths/values and ASQ. If PHQ-9 is >=8 they will get follow-up questions and SMFQ. Teens will get follow-up text message robot dialogues with topic based on if a referral was accepted and other priorities. Chats may encourage strengths and provide resources, goals, mindfulness apps, journaling or depression-Cognitive Behavior Therapy dialogues for PHQ positive teens. Parents: get resources. PCPs: will use TDM results and decision support to detect, educate on depression, and motivate for intervention. They earn MOC.

Follow Up Measures: All teens and parents: get email/text reminders to do questionnaires 3, 6 and 11.5 months (pre next HSV) after initial HSV. Teens positive on initial PHQ-9 in both groups will be paid (and called) to do a repeat PHQ-9 with follow-up about interval treatment and parents will do SMFQ and provide impressions of PCP management and success of any referrals. Rates for Ask Suicide Screening Questions (ASSQ) will be in the intervention group only, as it is not usual care, but any PCP may use it. Evaluation will include: depression screening rates, decision support use, proportions of positive teens referred via care coordination and teen use of resources.

II.7 Analysis of Results of Intervention: Initial: Descriptive analyses. Primary Questions 1&2: t-tests adjusted for design effect, categorical statistical tests of inference appropriately matched to the underlying distributions of the measures used at T1 and T2, adjusted for design. Secondary Question 2: Chi-Squared Test of Independence on two cross-sectional samples tabulated at T0 and T1. Rates of ASQ use will be assessed for T2-T3. Tests will be applied to 2 cross-sectional samples regardless of treatment arm. Multi-Level Linear Regression models for Primary Questions 1-2 and Logistic Regression models for Secondary Questions 1-3 will assess impact of patient characteristics and item responses, and control for design effect of a cluster-randomized design.

ELIGIBILITY:
Inclusion Criteria:

* English speaking teens
* English speaking caregivers

Exclusion Criteria:

* Non English speaking teens
* Non English speaking caregivers

Ages: 12 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: All teens coming to participating PCPs for well child visits during the study period and their adult caregivers for those under 18
Sampling Method: Probability Sample
Enrollment: 580 (Estimated)
Dates: Start 2021-02-01 (Actual); Primary Completion 2023-06 (Estimated); Study Completion 2023-06 (Estimated)

PRIMARY OUTCOMES:
Change in Short Moods and Feelings Questionnaire | Day 1 well visit, day 1 + 3 months, day 1 + 6 months, and day 1 + 11.5 months
  A brief screen of depressed mood completed by teen, 0-26 with 26 worst
Change in Short Moods and Feelings Questionnaire- Parent version | Day 1 well visit, day 1 + 3 months, day 1 + 6 months, and day 1 + 11.5 months
  A brief screen of depressed mood completed by parent, 0-26 with 26 worst

SECONDARY OUTCOMES:
Change in Self report of treatment access | Day 1 well visit when there is a positive depression screen, day 1 + 3 months, day 1 + 6 months, and day 1 + 11.5 months
  Teen report of depression treatment access, accessed or not accessed with accessed considered better
Patient Health Questionnaire-9 (PHQ-9) | Entire study period of up to 3 years
  Numbers of teens screened with PHQ-9 for depression. This outcome is not the score of the tool but numbers completing the tool with range 0-2600 with higher better.
Ask Suicide Screening Questions (ASSQ) | Entire study period of up to 3 years
  Numbers of teens screened with ASSQ for suicidal ideation, scores 0-8 with higher worst. This Outcome is number screened with range 0-2600 with higher better.

CONTACTS AND LOCATIONS:
Overall Officials: Barbara J Howard, MD, Principal Investigator — Total Child Health; Raymond A Sturner, MD, Principal Investigator — Center for Promotion of Child Development; Marianne Wamboldt, MD, Principal Investigator — U Colorado Medical Center
Locations (1):
- Total Child Health, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: Yes
After publication of results de-identified data may be available to qualified researchers.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Starting 6 months after results are published.
Access Criteria: Qualified medical or mental health researchers.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-02-05): https://cdn.clinicaltrials.gov/large-docs/85/NCT04489485/Prot_SAP_000.pdf